CLINICAL TRIAL: NCT04948944
Title: Frontal Stimulation to Modulate Threat Sensitivity in Anxious Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LIBR#2021-005; P20GM121312 (NIH)
Record Dates: First submitted 2021-03-12; First posted 2021-07-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Depression; Anxiety and Fear
Keywords: depression; anxiety; transcranial direct current stimulation; fMRI; startle reflex; threat sensitivity
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: treatment code provided by non-study staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active transcranial direct current stimulation (Experimental): The investigators use Soterix mini-CT Stimulator to deliver 30 minutes 2mAmp tDCS to the bilateral DLPFC (optimized lateral electrode placement montage), with the the anode on the left hemisphere and the cathode on the right hemisphere. The electrodes are rubber and are placed in an MRI compatible holder and affixed with conductive paste. The investigators will use a bespoke headstrap to place the electrodes, which are held in place by the conductive paste.
  Interventions: Device: transcranial direct current stimulation
- sham transcranial direct current stimulation (Sham Comparator): In the sham stimulation mode, the device shows pseudorandom numbers on the screen that look like real stimulation is being delivered. The device gives a low level of stimulation at the very beginning and at the very end of the stimulation session (30 seconds ramp up and 30 seconds ramp down) in order to recreate the feeling of tingling that subjects perceive at the beginning and end of real stimulation.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — the tDCS stimulator delivers very low (2mAmp) current with surface electrodes to the skull

SUMMARY:
Over 50% of patients with major depressive disorder (MDD) do not respond to initial treatment and relapse is common. In particular, comorbid depression and anxiety disorders are associated with more treatment resistance. Thus, there is a great need for novel, more targeted treatments. Transcranial direct current stimulation (tDCS) is a novel intervention that can be used to causally target neural excitability and plasticity in brain regions/circuits implicated in regulating mood and anxiety and emerging evidence suggests that it reduces threat sensitivity. Here the investigators propose to use tDCS to target threat sensitivity as a core symptom of anxious depression to determine if the investigators can engage the neural circuits that are treatment targets. Following the administration of a single dose of anxiolytic or antidepressant treatment, early changes in emotional processing have been observed in healthy people and clinical groups. Among patients, acute cognitive effects - such as a reduction in threat sensitivity - have been shown to predict response to drug and behavioral treatments. Functional magnetic resonance imaging (fMRI) studies have confirmed hyperactive amygdala and/or hypoactive prefrontal activity in patients, indicating an imbalance of activity within this cortico-limbic circuit that sub-serves threat identification (amygdala) and top-down control (prefrontal). Specifically, treatments aiming to remediate prefrontal/ amygdala dysfunction could be a critical target in patients exhibiting these deficits. Several clinical trials have shown that administration of frontal cortex tDCS is a potentially effective treatment for MDD. However, underlying mechanisms of action are unclear. To meet this gap, the investigators propose an experimental medicine study (target identification and initial target engagement paths) where 141 volunteers with anxious MDD will be randomized to receive a single session of active or sham tDCS in a parallel design. Threat sensitivity will be measured using task and resting state fMRI and potentiated startle electrophysiology. Preliminary data suggest reductions in behavioral threat sensitivity from a single session of frontal tDCS. This was followed up with an fMRI study which found that a single session of active vs sham frontal tDCS reduced amygdala response to fearful faces whilst simultaneously increasing frontal attentional control signals. This provides evidence that modulating activity in the frontal cortex inhibits amygdala response to threat, highlighting a potential neural mechanism for the behavioral reduction in threat sensitivity. In addition, this offers initial mechanistic insights into the efficacy of tDCS in clinical trials for the treatment of MDD and anxiety disorders, suggesting that threat sensitivity may be a suitable cognitive target. The current proposal builds on this to establish acute effects of frontal tDCS on amygdala response to threat (primary aim), frontoparietal response to threat (secondary aim), startle response under threat (secondary aim) and approach-avoidance-conflict (exploratory aim). The ultimate aim is to apply these multi-level acute findings to mechanistic clinical trials of tDCS, to test their prediction of treatment response (full model path) and improve patient outcomes.

DETAILED DESCRIPTION:
141 participants with anxious MDD were recruited from the community. Participants will undergo screening and baseline assessments using self-report and clinical assessments. Eligible participants will be invited for an additional screening session where they will allocated to either active or sham stimulation arms (50% in each arm). Participants in the active arm will receive 30 minutes tDCS over bilateral prefrontal cortex using an optimized lateral electrode (OLE) placement montage. This montage is selected as it is commonly used in clinical trials of tDCS for MDD and is designed to target the lateral DLPFC. Moreover, hypoactive frontal activation and related impaired top-down control is associated with MDD and anxiety disorders. Resting state (rs) fMRI data will be collected immediately before, during and after active or sham tDCS. After tDCS, task-based fMRI data (attentional control task with fearful distractors) and behavioral data (approach avoidance task) will be acquired. Mood will be assessed with a single item 0-100 visual analogue scale (VAS) question and Positive and Negative Affective schedule (PANAS) at multiple time points before and after imaging and tDCS. Subjective and neural responses to fearful faces in prefrontal cortical areas and subcortical-limbic areas (fearful>neutral) and their connectivity during resting state will be assessed with contrasts made between active and sham stimulation. Anxiety (unpredictable shock > neutral) and fear (predictable shock > neutral) potentiated startle will be measured using EMG. For additional exploratory analyses relating to blood based markers of neuroplasticity (Kynurenine), a blood sample will be taken.

ELIGIBILITY:
Inclusion criteria:

1. Current major depressive episode assessed by clinician administered MINI;
2. Minimum score of 8 on OASIS anxiety scale;
3. Normal or corrected to normal vision/hearing, as protocol elements may not be valid otherwise;
4. Fluent English speaker, capable of providing written informed consent

Exclusion criteria:

1. Has uncontrolled, clinically significant neurologic (including seizure disorders): cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results;
2. History of moderate or severe traumatic brain injury, as assessed by the Tulsa Head Injury Screen (THIS) questionnaire;
3. Family history of psychotic or bipolar disorder;
4. Current diagnosis of eating disorder or obsessive-compulsive disorder;
5. Current use of medications with major effects on the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, excessive caffeine intake > 1000 mg/day);
6. Moderate or severe current substance use disorder according to DSM 5 criteria, assessed via MINI;
7. Drug or alcohol intoxication (based on positive urine test or breathalyzer test at screen or baseline) or reported acute alcohol or drug withdrawal;
8. Has a risk of suicide according to the Investigator's clinical judgment or per Columbia-Suicide Severity Rating Scale (C-SSRS), the subject scores "yes" on items 4 or 5 in the Suicidal Ideation section with referent to a 30-day period prior to Screening/Baseline or the subject has had one or more suicidal attempts with reference to a 2-year period prior to Screening/Baseline;
9. MRI or tDCS contraindications;
10. Is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during this time-period;
11. History of highly irritable skin and/or contact dermatitis that affects skin integrity of the scalp;
12. Any participant judged by the Investigator to be inappropriate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
The difference between amygdala Blood-Oxygen-Level-Dependent (BOLD) functional Magnetic Resonance Imaging (fMRI) activation to fearful faces compared to neutral faces | immediately after intervention
  Preliminary findings show that frontal tDCS can reduce amygdala threat reactivity in high trait anxious females. The investigators seek to replicate this effect in a larger, clinical sample which also includes males. Specifically, the investigators expect that, compared to sham tDCS, the active tDCS group will show changed amygdala BOLD fMRI activation to fearful faces (difference between fearful and neutral faces), following acute tDCS administration.

SECONDARY OUTCOMES:
The difference between frontoparietal Blood-Oxygen-Level-Dependent (BOLD) functional Magnetic Resonance Imaging (fMRI) activation to fearful faces compared to neutral faces | immediately after intervention
  Preliminary findings show that frontal tDCS can increase frontoparietal activation to threat in high trait anxious females. The investigators seek to replicate this effect in a larger, clinical sample which also includes males. Specifically, the investigators expect that, compared to sham tDCS, the active tDCS group will show changed frontoparietal BOLD activation to fearful faces (difference between fearful and neutral faces), following acute tDCS administration.
The difference between startle reflex measured by electromyography (EMG) under threat of unpredictable shock compared to no threat of shock | immediately after intervention
  The significant acute reduction in behavioral threat sensitivity from a single session of tDCS is similar that seen with anxiolytic treatments. Anxiolytic treatments also reliably reduce startle response to unpredictable threat. The investigators hypothesize that compared to sham tDCS, the active tDCS group will show changed anxiety potentiated startle EMG (unpredictable shock minus no shock condition) following acute tDCS administration.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ironside, DPhil, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT04948944/Prot_ICF_000.pdf